CLINICAL TRIAL: NCT05044377
Title: Study on Optimal Treatment Strategy for Elderly Patients With High-risk Complex Aortic Valve Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yongjian Wu (Other Government)
Responsible Party: Sponsor-Investigator, Yongjian Wu, Chief physician, China National Center for Cardiovascular Diseases
Organization: China National Center for Cardiovascular Diseases (Other Government)
Other Study IDs: high-risk AS 2020-08
Record Dates: First submitted 2021-09-12; First posted 2021-09-14 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aortic valve disease (AVD) is the most common and age-related mortality in elderly patients with valvular heart disease (VHD). Although transcatheter aortic valve replacement (TAVR) has been recommended at a higher level in foreign guidelines, there are still many high-risk and severe elderly patients with VHD who have not received effective treatment because of many complications and untimely medical treatment. Different from Europe and the United States, the majority of patients with bicuspid aortic valve are in China, and the calcification is more serious. The current clinical evaluation system and treatment guidelines can not be effectively applied to the high-risk and complex elderly patients. Therefore, the investigators should train and set up a valvular heart disease team, explore the technical difficulties of TAVR treatment in such patients, establish emergency TAVR operation mechanism, build a clinical evaluation system for high-risk and complex elderly patients with aortic valve disease in China, evaluate the curative effect periodically and further optimize the treatment strategy, so as to improve the quality of life and the meaning of life cycle of elderly patients with VHD in China Great significance.

ELIGIBILITY:
Inclusion Criteria:

* • patients over 75 years old meet one of the following conditions. severe valvular heart disease as defined by echocardiography:

  1. aortic stenosis, moderate or above, or valve area ≤1.0cm2, or maximal jet velocity ≥4.0m/sec, or mean pressure gradient ≥40mmHg,
  2. aortic regurgitation, moderate or above, or jet width ≥65% of left ventricular outflow tract, or regurgitant volume≥60ml/beat, or regurgitant fraction ≥50%,

Exclusion Criteria:

* • Patients cannot be followed up for any reasons.
* •Patients have been enrolled in this study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Seven cooperative hospitals with cardiovascular as the key specialty in Beijing have continuously registered patients with severe aortic valve disease aged 75 years or older.
Sampling Method: Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 1 year
  The primary endpoint of this study is 1 years all-cause mortality all stroke and re-hospitalization (for valve-related decompensation or procedure-related complications) .

CONTACTS AND LOCATIONS:
Overall Officials: yongjian wu, doctor, Study Chair — Fuwai Hospital, National Center for Cardiovascular Diseases，Chinese Academy of Medical Sciences
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No